CLINICAL TRIAL: NCT04317209
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study on Safety, Tolerability and Pharmacokinetics of SHR0410 in Hemodialysis Subjects With Moderate to Severe Pruritus
Brief Title: A Study of SHR0410 in Hemodialysis Patients With Pruritus
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR0410-103
Record Dates: First submitted 2020-03-16; First posted 2020-03-23 (Actual); Last update posted 2020-05-22 (Actual); Status verified 2020-05

CONDITIONS: Pruritus
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SHR0410 low dosage (Experimental)
  Interventions: Drug: SHR0410
- SHR0410 medium dosage (Experimental)
  Interventions: Drug: SHR0410
- SHR0410 high dosage (Experimental)
  Interventions: Drug: SHR0410
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SHR0410 — administered intravenously
  Other Names: KOR agonist
  Arms: SHR0410 high dosage; SHR0410 low dosage; SHR0410 medium dosage
Drug: Placebo — administered intravenously
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the safety, tolerability and pharmacokinetics of SHR0410 in hemodialysis patients with moderate to severe pruritus

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18-65 (inclusive);
2. Weight (> 50 kg);
3. Patients with end-stage renal disease receiving hemodialysis (including hemodialysis and hemofiltration) three times a week for at least 3 months.
4. VAS≥4 at screening

Exclusion Criteria:

1. New York cardiac function classification (NYHA) ≥ level III in the current or previous 6 months;
2. Pruritus caused by other than end-stage renal disease or its complications..
3. History of malignancy
4. Any physical or mental illness or condition, as determined by the study investigator, that may increase the risk of participating the trial, affect the subject's compliance with the protocol, or affect the subject's completion of the trial
5. Positive urine drug screening; Or a history of drug abuse;
6. Urine test positive for nicotine;
7. Alcohol breath test positive;
8. Alanine aminotransferase (ALT), aspartate aminotransferase (AST) or transglutaminase (GGT) was 1.5 times higher than the upper limit of normal value (ULN), or total bilirubin was 1.5 times higher than the upper limit of normal value (ULN);
9. Screening for hepatitis c antibody (HCVAb), syphilis antibody or human immunodeficiency virus (HIV) antibody positive; Or hepatitis B is active;
10. Abnormal electrocardiogram considered inappropriate to participate in this study by the investigator
11. positive for human chorionic gonadotropin (hCG) blood test
12. A history of allergies to opioids
13. Has used opioids within one week prior to the current visit, or cannot avoid to use opioids other than the study drug during the study period;
14. Change the treatment regimen for pruritus within 14 days, or cannot avoid to change the treatment regimen for pruritus during the study period
15. Received Ultraviolet phototherapy within 14 days before screening visit; Or cannot avoid to receive ultraviolet light therapy during the study.
16. Change the treatment regimen of gabapentin, pregabalin, or duloxetine within 14 days before screening visit; Or the treatment regimen of gabapentin, pregabalin, or duloxetine cannot be avoided to be changed during the study period.
17. Change the treatment regimen of medications within 14 days that may affect the judgment of antipruritic effect; Or the treatment regimen cannot be avoided to be changed during the study
18. Using topical antipruritic drugs, such as creams and patches with moisturizing or antipruritic effects at present.
19. Kidney transplantation is expected during the study period;
20. Subjects who had Participated in this trial (defined by signing the informed consent);
21. Subjects who had Participated in clinical trials of any other drugs within the previous 3 months; Or plan to participate in other drug trials during the trial period;
22. Subjects who had Participated in the clinical trial of any medical device within the previous 3 months; Or participate in other medical device tests during the trial period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2020-05-17 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of any adverse events that occurred between the first administration and the 48-hour period following the last administration | up to 7 days
  To evaluate the safety and tolerability of repeated doses of SHR0410

SECONDARY OUTCOMES:
Area under drug-time curve | up to 7 days
  To evaluate pharmacokinetic (PK) of repeated doses of SHR0410
peak time | up to 7 days
  To evaluate pharmacokinetic (PK) of repeated doses of SHR0410
peak concentration | up to 7 days
  To evaluate pharmacokinetic (PK) of repeated doses of SHR0410
half-life | up to 7 days
  To evaluate pharmacokinetic (PK) of repeated doses of SHR0410
apparent clearance rate | up to 7 days
  To evaluate pharmacokinetic (PK) of repeated doses of SHR0410
apparent distribution volume | up to 7 days
  To evaluate pharmacokinetic (PK) of repeated doses of SHR0410
The ratio of AUC0-t after the first and last administration. | up to 7 days
  To evaluate pharmacokinetic (PK) of repeated doses of SHR0410

CONTACTS AND LOCATIONS:
Locations (1):
- The first affiliated hospital of sun yat-sen university, Guangzhou, China

IPD SHARING:
Plan to Share IPD: No